CLINICAL TRIAL: NCT02362139
Title: The Impact of Papaverine on First Stage of Labor
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: eran ashwal (Other)
Responsible Party: Sponsor-Investigator, eran ashwal, doctor, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0463-13-RMC
Record Dates: First submitted 2015-02-08; First posted 2015-02-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Duration of Labor.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The study group (Experimental): 200 pregnant women, 18-45 years old, 37-41 weeks of gestation, in spontaneous labor, which were treated with 80 mg of Intra-muscular (IM) Papverine during the latent phase of labor (cervical dilatation<4cm).
  Interventions: Drug: The study group
- The control group (No Intervention): 200 pregnant women, 18-45 years old, 37-41 weeks of gestation, in spontaneous labor, which were not treated with IM Papverine

INTERVENTIONS:
Drug: The study group — 200 pregnant women, 18-45 years old, 37-41 weeks of gestation, in spontaneous labor, which were treated with 80 mg of Intra-muscular (IM) Papverine during the latent phase of labor (cervical dilatation<4cm).
  Other Names: Papverine
  Arms: The study group

SUMMARY:
In the investigators institution, there is a wide use of Papaverine in delivery room, but this use is optional, and is left to the discretion of the physician.

The aim of the investigators study is to prospectively evaluate the influence of Papaverine administration in the latent phase of labor, on the duration of labor.

DETAILED DESCRIPTION:
Cervical dilatation rate and the duration of delivery are key issues in the management of labor. Protracted labor is known to be associated with a range of potential maternal and neonatal complications, including higher rate of post partum hemorrhage (PPH), cesarean sections, instrumental deliveries, maternal or neonatal infections and neonatal pulmonary asphyxia [1,2,3]. Thus, there is a rationale for reducing the duration of labor in order to reduce adverse pregnancy outcome.

Active management of labor as was demonstrated by O'driscoll et al. was found to be effective in shortening the duration of delivery [1, 4]. There is a variety of mechanical and medical methods for labor induction and augmentation. Mechanical methods include artificial rupture of membranes (amniotomy), with or without the use of Pitocin [5, 6], manual sweeping of the amniotic membranes which promotes the release of prostaglandins [7], and extra-amniotic balloon [8]. Medical methods such as prostaglandins and Pitocin are well studied and were found to reduce the duration of labor.

Papaverine and its derivatives have been studied in the nineties of the last century and were found to be effective in reducing the duration of the first stage of labor [9, 10, 11]. Drotaverine hydrochloride is an analog of Papaverine and a selective inhibitor of phosphodiesterase 4. It was found to be effective in accelerating cervical dilatation through smooth muscle relaxation.

In a prospective randomized controlled trial that included 146 women in spontaneous vaginal delivery, Madhu et al. have shown that women who were treated with Drotaverine through the latent phase of labor, had significantly shorter duration of time between the administration of the medication and the delivery of the fetus, compared to women that were treated with placebo (182 minutes compared to 245 minutes with placebo). Moreover, the cervical dilatation rate in the Drotaverine group was significantly higher than this in the placebo group (3 centimeters per hour (cm\Hr) compared to 1.4 cm\Hr) [9]. These findings are in agreement with Shmara et al. that have also demonstrated a significant reduction in the duration of labor and a significant acceleration in cervical dilatation rate with Drotaverine administration compared to placebo. In this study 100% of women who were treated with Drotaverine in the latent phase of labor have delivered in 6 hours from the administration, compared to 46% in the placebo group [10].

Only few previous studies have addressed the influence of Papaverine administration on the duration of labor [9-12], and these studies are limited by small sample size, and different administration protocols. Moreover, in part of these studies, the use of Papaverine was not separate from the use of other methods for labor augmentation such as amniotomy or Pitocin administration, what could bias their results.

In the investigators institution, there is a wide use of Papaverine in delivery room, but this use is optional, and is left to the discretion of the physician.

The aim of the investigators study is to prospectively evaluate the influence of Papaverine administration in the latent phase of labor, on the duration of labor.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy.
* 37-41 weeks of gestation.
* Women who enter delivery room in spontaneous labor during the latent phase of labor (cervical dilatation <4cm).
* Maternal age between 18 and 45.

Exclusion Criteria:

* Women who enter delivery room during the active phase of labor (cervical dilatation greater than 5 cm).
* Women with previous cesarean section
* Women with premature rupture of membranes (PROM)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
The duration of time between Papaverine administration and delivery. | 24 month

SECONDARY OUTCOMES:
Duration of second and third stages of labor | 24 month
Cervical dilatation rate (cm\Hr) | 24 month
Papaverine adverse outcome | 24 month
  Papaverine Side effects: nausea and vomiting, palpitations, maternal tachycardia (>100 BpM), neonatal tachycardia (base line> 160 BpM for 10 minutes or more), headache.
  o Monitoring for side effects will be performed every hour

CONTACTS AND LOCATIONS:
Overall Officials: Eran Ashwal, MD, Principal Investigator — Rabin Medical Center